CLINICAL TRIAL: NCT06028841
Title: An Open-label Phase 3 Trial to Assess the Safety and Immunogenicity of a Live-attenuated Chikungunya Virus Vaccine (VLA1553) in Moderately Immunocompromised Adult Participants Infected with Human Immunodeficiency Virus
Brief Title: A Clinical Phase 3 Trial of VLA1553 in Adult Participants with Human Immunodeficiency Virus (HIV)
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Withdrawn due to challenges related to recruitment.
Sponsor: Valneva Austria GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: VLA1553-304
Record Dates: First submitted 2023-03-29; First posted 2023-09-08 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Chikungunya Virus Infection
MeSH Terms: conditions — Chikungunya Fever

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- VLA1553 (Experimental)
  Interventions: Biological: VLA1553

INTERVENTIONS:
Biological: VLA1553 — Single intramuscular vaccination on Day 1 with VLA1553, a lyophilized live-attenuated Chikungunya vaccine candidate 1x10E4 TCID50 per dose

SUMMARY:
This was a phase 3 clinical study to evaluate the safety, tolerability, and immunogenicity of VLA1553 in moderately immunocompromised adults with HIV infection.

DETAILED DESCRIPTION:
This was a multicenter, prospective, open-label, uncontrolled, single arm, phase 3 clinical study evaluating the final dose of VLA1553. The safety, tolerability, and immunogenicity of VLA1553 should have been assessed in moderately immunocompromised adult participants infected with HIV living in CHIKV endemic areas. Approximately 75 male and female adults (aged 18 years or above) infected with HIV should have been enrolled. Participants would have been screened by ELISA for evidence of previous CHIKV exposure excluding CHIKV seropositive participants from study participation.

ELIGIBILITY:
Inclusion Criteria:

Participants who met ALL of the following criteria were eligible for this study:

1. Adult participant aged 18 years or above infected with HIV of either gender
2. Participant has an understanding of the study and its procedures, agrees to its provisions, and voluntarily gives written informed consent prior to any study-related procedures
3. Stage of disease A1, A2, B1 or B2 according to the revised CDC classification system for HIV infection from 1993 or Stages 1 or 2 in the absence of AIDS defining conditions (CDC update from 1994)
4. Participants are recruited in Cohorts:

   1. For Cohort I:

      Participant has CD4+ T cell counts >350-≤400 cells/μL, is receiving antiretroviral therapy (ART) for at least 6 months and plasma HIV RNA < 400 copies/ mL prior enrollment
   2. For Cohort II:

   Participant has CD4+ T cell counts >200 cells/μL (no upper limit), is receiving ART for at least 3 months and plasma HIV RNA < 50 copies/ mL prior enrollment
5. Participant is seronegative for previous CHIKV exposure (i.e. IgM- and IgG-) as screened by CHIKV-specific ELISA
6. If female participant is of childbearing potential:

   1. Participant has a negative urine pregnancy test at screening (Visit 0) or Day 1 (Visit 1), respectively
   2. Participant has practiced an adequate method of contraception during the 30 days before screening (Visit 0)
   3. Participant agrees to employ adequate birth control measures for the first three months post-vaccination (i.e. until Day 85, Visit 6).
7. Female/male participant agrees to employ adequate birth control measures for the first three months post-vaccination (i.e., until Day 85, Visit 7)

Exclusion Criteria:

Participants who met ANY of the following criteria were NOT eligible for this study:

1. Participant is taking medication or other treatment for unresolved symptoms attributed to a previous CHIKV infection; or has participated in a clinical study involving an investigational CHIKV vaccine
2. Participant has an acute or recent infection (and who is not symptom-free in the week prior to the Screening Visit (Visit 0) and Visit 1)
3. Participant tests positive for human immunodeficiency virus (HIV) and fulfills AIDS indicator T cell counts or AIDS indicator conditions (disease stages C1, C2 or C3 or stage
4. Participant tests positive for HIV with the actual target disease stages A1, A2, B1 or B2 (or stage 1 or 2), but was classified in the past at least once as fulfilling AIDS indicator conditions (disease stage C1, C2 or C3) or AIDS indicator T cell counts (CD4+ lymphocyte count <200/μL or CD4+ percentage <14%)
5. Participant tests PCR positive for active hepatitis B or hepatitis C virus (HCV)
6. Participant has received any vaccine within 28 days prior to vaccination in this study or plans to receive any vaccine within 28 days after vaccination
7. Participant has abnormal findings in any required study investigations (e.g. medical history, physical examination, and laboratory findings) considered clinically relevant by the Investigator and which pose a risk for participation in the study based on his/her judgement
8. Participant currently has or had a history of significant cardiovascular, respiratory, metabolic, neurological, hepatic, rheumatic, autoimmune, hematological, gastrointestinal or renal disorder (of note: Mild asthma that requires low dose corticosteroid inhalation only, during limited time periods of the year is not an exclusion criterion)
9. Participant has an abnormal, clinically significant 12-lead ECG at screening
10. Participant has a history of immune-mediated or clinically relevant arthritis/arthralgia
11. Participant has a history of malignancy
12. Participant has a known or suspected defect of the immune system that can be expected to influence the immune response to the vaccine other than asymptomatic or moderately symptomatic HIV infection, such as participants with congenital immunodeficiency, status post organ transplantation or immuno-suppressive therapy within four weeks prior to Visit 1. Immuno-suppressive therapy is defined as administration of chronic (longer than 14 days) prednisone or equivalent ≥0.05 mg/kg/day within 4 weeks prior to study entry, radiation therapy or immunosuppressive cytotoxic drugs/ monoclonal antibodies in the previous three years; topical and inhaled steroids are allowed
13. Participant has a history of any vaccine related contraindicating event (e.g., anaphylaxis, allergy to components of the candidate vaccine, other known contraindications including febrile convulsions)
14. Participant presents with clinical conditions representing a contraindication to intramuscular vaccination and blood draws
15. Participant is pregnant (positive urine pregnancy test at screening or Visit 1, respectively), is lactating at the time of enrollment, has plans to become pregnant or subject's female partner plans to become pregnant during the first three months post-vaccination or practices unreliable contraception
16. Participant received blood-derived products (e.g. plasma) within 90 days prior to vaccination in this study
17. Participant has a rash, dermatological condition or tattoos that would, in the opinion of the Investigator, interfere with injection site reaction rating
18. Participant has participated in another clinical study involving an investigational medicinal product (IMP) or device within 30 days prior to vaccination or is scheduled to participate in another clinical study involving an IMP, or device during the course of this study
19. Participant is a member of the team conducting the study or in a dependent relationship with one of the study team members. Dependent relationships include close relatives (i.e., children, partner/spouse, siblings, parents) as well as employees of the Investigator or site personnel conducting the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-04-10 (Actual); Primary Completion 2024-08-27 (Actual); Study Completion 2024-08-27 (Actual)

PRIMARY OUTCOMES:
Solicited adverse events | until Day 15
To assess frequency and severity of unsolicited AEs | until Day 29 and Day 180 post-vaccination
To assess frequency and relatedness of any serious adverse event (SAE) | until Day 180 post-vaccination
To assess frequency and severity of any early onset adverse event of special interest (AESI) | within 2 to 21 days post-vaccination (i.e. Day 3 - Day 22)
To assess frequency and severity of any late onset adverse event of special interest (AESI) during the entire study | starting 22 days post-vaccination (i.e. Day 23 - Day 180)
To assess CHIKV viremia | on Days 1, 4, 8 and 15 (Day 29 and Day 57, if applicable)
To assess HIV viral load | on Days 1, 15, 29, 57, 85, and 180

SECONDARY OUTCOMES:
Immune response as measured by CHIKV-specific neutralizing antibody titers post-vaccination as determined by μPRNT assay | Day 15, Day 29, Day 57, Day 85 and Day 180
Proportion of participants with seroresponse levels post-vaccination as determined by μPRNT assay | Day 15, Day 29, Day 57, Day 85 and Day 180
Proportion of participants with seroconversion as compared to baseline as determined by μPRNT assay | Day 29 and Day 180
Fold increase of CHIKV-specific neutralizing antibody titers determined by μPRNT assay post-vaccination as compared to baseline | Day 15, Day 29, Day 57, Day 85 and Day 180
Proportion of participants reaching an at least 4-fold, 8-fold, 16-fold or 64-fold increase in CHIKV-specific neutralizing antibody titer compared to baseline as measured by μPRNT assay | Day 15, Day 29, Day 57, Day 85 and Day 180

CONTACTS AND LOCATIONS:
Overall Officials: Valneva Clinical Development, Study Chair — Valneva Austria GmbH

IPD SHARING:
Plan to Share IPD: Undecided